CLINICAL TRIAL: NCT07324252
Title: Feasibility of Small RNA Profiling by Next-Generation Sequencing in Exhaled Breath Condensate and Its Modulation by Maximal Exercise: a Pilot Study
Brief Title: Small RNA Profiling in EBC in Athletes
Acronym: AirBiopsy
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lukasz Minarowski, Head of Department of Respiratory Physiopathology, Medical University of Bialystok
Other Study IDs: APK.002.584.2024; B.SUB.25.512 (Other: Medical University of Bialystok)
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Exhaled Breath Condensate; Athlete; RNA Profile; Cardio-pulmonary Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 22 EBC samples collected with the RTube device from 11 healthy volunteers and 3 patients with lung cancer and co-existing COPD (GOLD 3-4), at rest and after standardised maximal exercise confirmed by cardiopulmonary exercise testing (CPET). Total RNA was extracted using a commercial high-throughput RNA isolation kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exhaled breath condensate donors: athletes (22) and lung cancer (3) donors of EBC

SUMMARY:
Background: Exhaled breath condensate (EBC) is a non-invasively collected biofluid containing volatile and non-volatile compounds, including small RNAs. Small RNA profiling in EBC appears to be a promising approach for identifying and developing minimally invasive biomarkers for lung diseases; however, methodological evidence remains limited and heterogeneous.

Objectives: To evaluate the technical feasibility of small RNA extraction and next-generation sequencing (NGS) from EBC and to characterise small RNA profiles at rest and after maximal exercise, using EBC as a model matrix for dynamic physiological changes.

Methods: In a pilot study conducted as part of statutory research at the Medical University of Białystok (B.SUB.25.512 and B.SUB.25.529), we analysed 22 EBC samples collected with the RTube device from 11 healthy volunteers and 3 patients with lung cancer and co-existing COPD (GOLD 3-4), at rest and after standardised maximal exercise confirmed by cardiopulmonary exercise testing (CPET). Total RNA was extracted using a commercial high-throughput RNA isolation kit designed for biological samples with low nucleic acid content, the miRNeasy Serum/Plasma Advanced Kit (Qiagen), according to the manufacturer's protocol with modifications. Small RNA libraries were generated using the high-sensitivity, low-input TrueQuant Small RNA-Seq Library Preparation Kit (GenXPro GmbH) with Unique Molecular Identifiers (UMIs) and sequenced on an Illumina platform. Reads were processed with Cutadapt and FastQC, mapped iteratively to the hg38 (Homo sapiens) reference genome using Bowtie2, aligned against an array of RNA databases, including miRNA (miRBase), tRNA (GtRNAdb), piRNA (piRNAdb), ncRNA (ENSEMBL), and cDNA (ENSEMBL) and quantified with HTSeq. Differential expression analysis (DEA) and principal component analysis (PCA) were performed with DESeq2.

ELIGIBILITY:
Inclusion Criteria:

* ability to perform CPET
* ability to perform spirometry

Exclusion Criteria:

* lack of informed consent
* absolute contradictions to CPET or spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volouteers, amateur athletes (runners) and lung cancer patients with stage IIIb or VI disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
smallRNA profile | From August 2025 to December 2025
EBC collection | From January 2025 to August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Physiopathology, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
detailed RNA profile and clinical data available on demand
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026 to January 2027
Access Criteria: researchers and interested parties after an assessment of the data usage description and appropriate bioethical agreement